CLINICAL TRIAL: NCT05044299
Title: Development of the Isoped Device for Increasing Blood Flow in a Sedentary Aging Population
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The project was not considered for funding so we scrapped the project.
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, David Bradshaw, Adjunct research assistant professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IsopedPhase1
Record Dates: First submitted 2021-09-01; First posted 2021-09-14 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Sedentary Behavior; Aging
Keywords: aging; sedentary behavior; blood flow; device
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Study has two arms comparing device with and without resistance load over equal period of operation
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isoped mobilization with resistance load (Active Comparator): Use of Isoped with movement at 3 levels of resistance load: zero, low, high, each condition lasts 3 minutes at 9 minutes total work
  Interventions: Device: Isoped
- Isoped mobilization without resistance load (Active Comparator): Use of Isoped with movement at zero resistance load lasts 9 minutes of work
  Interventions: Device: Isoped

INTERVENTIONS:
Device: Isoped — Isoped is a mechanical device allowing movement of lower extremities in a forward and backward motion, with phone-based app to control resistance load

SUMMARY:
The Isoped (patented) is a portable medical device that provides a safe and engaging opportunity for regular physical activity to those with limited mobility and difficulties with performing traditional exercise tasks. It is a tool designed to encourage regular and repeated low impact movement of the lower extremities that can improve blood flow and lead to improved cardiovascular function. By restoring healthier cardiovascular tone, Isoped users may be able to progress to more demanding activities leading to a healthy lifestyle change. Experiencing these improvements can boost confidence, mood, and overall quality of life. Isoped users can exercise while sitting at a desk, watching television, or in a rehabilitation facility. The lightweight device sits on the floor beneath the user's feet and can be operated from a seated, reclined, or supine position. Circulation and lower extremities' blood flow increase as the feet slide the pedals in a forward and backward movement similar to a shuffling walk or in cross-country skiing. Resistance load can be controlled by the user for a customized experience using a smartphone app. Physical exercise is widely recommended as a primary treatment by physicians to improve circulation and prevent cardiovascular diseases associated with physical inactivity and a sedentary lifestyle. Isoped is a healthy and innovative alternative to pharmacological, surgical or other treatment modalities.

DETAILED DESCRIPTION:
Aim 1, Refine Device Prototype: A prototype Isoped device will be refined and calibrated for use. Engineering challenges include refining the design to incorporate these features and functions: Electronic Resistance mode (adjustable wirelessly through the Graphical User Interface (GUI)); Stride Length Adjustment (through the GUI); Stride Width Adjustment; Incline Adjustment (powered or manual); Footpad rotation and removal; Bluetooth connectivity to the GUI; comfortable stabilizing modifications to footpads.

Aim 2, Evaluate Device Efficacy and Safety: Isoped will be evaluated for safety and efficacy in a pilot clinical study of 40 volunteers aged 65 to 85 meeting criteria for a sedentary lifestyle and limited physical activity. To non-invasively determine the peripheral hemodynamic effect of the Isoped, we will quantify the lower extremity blood flow response to Isoped facilitated lower leg movement using doppler ultrasound measured at the femoral artery. Changes in mean blood pressure and heart rate will provide secondary measures of effect. Participant safety will be monitored using a 12-lead ECG and beat-by-beat measures of blood pressure and cardiac output. Device performance and safety will be evaluated by recording any deviations in device operability and any adverse events.

On completion of Phase 1, Phase 2 funding will provide the means to further evaluate the device for use in a patient population as a means for encouraging progression to regular health improving exercise regimens. A planned clinical trial in frail and sedentary aging persons using the Isoped over a period of several weeks will evaluate health improvement and willingness to engage in more demanding exercise regimens. This will position Isoped for commercialization as a tool for encouraging effective non-invasive, low-impact activity for improving the health and quality of life in a wide variety of patients having compromised circulation and who are unable and/or unwilling to engage in more rigorous physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported sedentary behavior and physically inactive
* Activity level confirmed via questionnaire
* Activity level confirmed by wearing activity monitor (Actigraph) over 7 days

Exclusion Criteria:

* History of cardiopulmonary
* History of cardiovascular pathology
* History of musculoskeletal conditions
* Other pathology precluding light exercise as evaluated by licensed geriatrician

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Blood flow | 15 minutes
  blood flow measured at femoral artery using doppler ultrasound

SECONDARY OUTCOMES:
continuous heart rate | 15 minutes
  heart rate measured using Finapres
continuous blood pressure | 15 minutes
  systolic, diastolic, and mean blood pressure measured continuously (Finapres)

CONTACTS AND LOCATIONS:
Overall Officials: David H Bradshaw, PhD, Principal Investigator — University of Utah

IPD SHARING:
Plan to Share IPD: No